CLINICAL TRIAL: NCT04798066
Title: Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of HB-adMSCs for the Treatment of Patients With Post-COVID-19 Syndrome
Brief Title: Intermediate Size Expanded Access Protocol for the Treatment of Post-COVID-19 Syndrome
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBPCOV01
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Post COVID-19 Syndrome
Keywords: Long Haul COVID-19; COVID-19; SARS-CoV-2; Long Haulers; Stem Cells; MSCs; Mesenchymal Stem Cells; COVID; Post COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: HB-adMSCs — Autologous adipose derived mesenchymal stem cells

SUMMARY:
This is an Intermediate- Size Patient Population Expanded Access Protocol to evaluate the safety and efficacy of HB-adMSCs for the treatment of patients with Post-COVID-19 Syndrome. The investigational product will be an add-on treatment to the standard of care.

DETAILED DESCRIPTION:
Visit 1 - Screening During the screening visit, the principal investigator and/or delegated staff must provide a copy of the IRB-approved informed consent form * to the subject before performing any study procedure.

* IRB must provide a certificate action as proof of approval of the informed consent form.

The study subject should take enough time to read this essential document. If the study subject agrees to participate in the clinical trial, after reading the document, he/she must sign it. By giving his/her signature, study subject allows the principal investigator and/or designated staff to perform the following study procedures:

1. Collection of medical history and demographic information.
2. Collection of prior (up to a week before screening) and current medications.
3. Evaluation of Inclusion and Exclusion Criteria.
4. Measurement of Weight in lb. and Height in inches.
5. Collection of vital signs, including respiratory rate, pulse rate, SPO2, blood pressure and body temperature.
6. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate, and urine pregnancy test if female of childbearing potential.
7. Completion of Patient Questionnaires, VAS of Symptom's and Fatigue Scale.
8. Physical Examination by the principal investigator.
9. Adverse Events Monitoring. Within a 28-day period, all screening data should be collected and analyzed, and the principal investigator must decide whether the screened subject is eligible to participate in this Intermediate- Size Patient Population Expanded Access Protocol.

Visit 2, 3, 4*, 5 and 6. (Infusions 1, 2, 3*, 4 and 5) Throughout these visits, the principal investigator and/or delegated staff will perform the following assessments:

1. Pre-Infusion Check List
2. Update Medical History Form if necessary.
3. Update Concomitant medications list if applicable. (no premedication necessary for the infusions)
4. Measurement of Weight in lb.
5. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
6. Completion VAS of Symptom's and Fatigue Scale.
7. Physical Examination by the principal investigator.
8. Investigational Product Administration:

   * Drug Name: HB-adMSCs
   * Route: Intravenous
   * Dose: 200 million.
9. 24 hours telephone encounter after Investigational Product Administration to assess incidence of adverse events or serious adverse events.
10. Adverse Events monitoring.

    * At Visit 4/Infusion 3: Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein, Erythrocyte sedimentation rate, urine pregnancy test female of childbearing potential and Patient Questionnaire.

Visit 7 (Follow up 1/Phone call)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Adverse Events monitoring.

Visit 8. (End of Study)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate, SPO2, blood pressure and body temperature.
5. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein, Erythrocyte sedimentation rate and urine pregnancy test if female of childbearing potential.
6. Completion of Patient Questionnaires, VAS of Symptom's and Fatigue Scale.
7. Physical Examination by the principal investigator.
8. Adverse Events monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 18-65 years at the time of signing the informed consent form.
2. Subject has had a positive SARS-COV-02 test (preferably PCR) within the last 12 months or has been diagnosed presumptive positive and has been treated for COVID-19 within the last 12 months.
3. Subject have not fully recovered from COVID-19 in weeks or months despite a negative Sars-COV-02 test and has been diagnosed with Post COVID-19 syndrome.
4. Subject is experiencing 2 or more symptoms for over 12 weeks either continually or intermittently with relapses not experienced pre-illness, that interferes with normal daily activities. Symptoms must be new symptoms, or dramatic worsening of symptoms i.e., subject didn't have symptoms, and had not sought medical treatment for the symptomsprior to COVID-19, or the symptoms are dramatically worse (in severity and frequency).

   * Extreme fatigue - feeling overtired with low energy and a strong desire to sleep.
   * Shortness of breath - (dyspnea) a feeling of being winded, difficulty in breathing, or a hunger for air.
   * Cough - hacking, or dry barking sound lingering dry or wet.
   * Brain fog -a diminished mental capacity marked by the inability to concentrate or to think or reason clearly that interferes with daily activities.
   * Headache - Sharp or dull reoccurring or intermittent that were not present pre-illness
   * Body aches - muscle soreness or generalized achiness throughout the body.
   * Joint pain - pain in the joints due to inflammation not experienced before illness.
   * Chest pain - (angina) feeling pressure, fullness, or tightness in your chest
   * Sleep issues - any sleep disturbances in sleep quality that makes sleep see inadequate or unrefreshing like insomnia or hypersomnia.
   * Loss of Taste/Smell - Diminished sense of taste or smell.
5. Subject must have previously banked their cells at Hope Biosciences, LLC.
6. Subject and sexual partner if woman of childbearing potential must use a least 1 highly effective form of birth control* throughout the study and for 6 months after the last dose of the investigational product.

(*Highly methods of birth control include, true sexual abstinence, bilateral tubal ligation, vasectomy, intrauterine. device and hormonal contraceptive methods.)

Exclusion Criteria:

1. Subject is unable to provide informed consent or to comply with study requirements.
2. Subject has currently been diagnosed with active COVID-19 disease.
3. Subjects unwilling to agree to the use of acceptable methods of contraception throughout the study and for 6 months after the last dose of the investigational product.
4. Pregnant or Breast-feeding women.
5. Subject has known alcoholic addiction or dependency, uses alcohol daily, or has current substance use or abuse.
6. Subject has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
7. Subject has 1 or more significant concurrent medical conditions (verified by medical records), including the following:

   * Poorly controlled diabetes mellitus (PCDM) defined as history of deficient standard of care treatment and/or pre-prandial glucose >130mg/dl during screening visit.
   * Medical History of Chronic kidney disease (CKD) diagnosis and/or screening results of eGFR < 59mL/min/1.73m2.
   * Presence of New York Heart Association (NYHA) Class III/IV heart failure during screening visit. (Appendices E)
   * Any medical history of myocardial infarction in any of the different types, such as ST-elevation myocardial infarction (STEMI) or non-ST-elevated myocardial infarction (NSTEMI), coronary spasm, or unstable angina.
   * Medical history of uncontrolled high blood pressure defined deficient standard of care treatment and/or blood pressure > 180/120 mm/Hg during screening visit.
   * Medical history of inherited thrombophilias, recent major general surgery, lower extremity paralysis due to spinal cord injury, fracture of the pelvis, hips, femur, cancer of the lung, brain, lymphoma, gynecologic system (ovary or uterus), or gastrointestinal tract (like pancreas or stomach).
8. Subject has received any stem cell treatment within 12 months before first dose of investigational product.
9. Subject has laboratory abnormalities during screening, including the following:

   * White blood cell count < 3000/mm3
   * Platelet count < 125,000mm3
   * Absolute neutrophil count < 1500/mm3
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN) x 1.5
   * Subject has any other laboratory abnormality, which, in the opinion of the investigator poses a safety risk or will prevent the subject for completing the study.
10. Subject is unlikely to complete the study or adhere to the study procedures.
11. Subject has a preexisting lung condition such as Chronic obstructive pulmonary disease (COPD).
12. Subjects with HIV, Hepatitis B and Hepatitis C.
13. Subject has a previously diagnosed psychiatric condition which in the opinion of the investigator may affect self-assessments.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

REFERENCES:
- [Result] Vij R, Kim H, Park H, Cheng T, Lotfi D, Chang D. Adipose-derived, autologous mesenchymal stem cell therapy for patients with post-COVID-19 syndrome: an intermediate-size expanded access program. Stem Cell Res Ther. 2023 Oct 5;14(1):287. doi: 10.1186/s13287-023-03522-1. PMID 37798650
- See also: Hope Biosciences LLC — https://www.hope.bio/
- See also: Hope Biosciences Stem Cell Research Foundation — https://www.hopebio.org/